CLINICAL TRIAL: NCT06264778
Title: Exploration of Fenestration Decompression Combined With Dalafenib in the Treatment of BRAF Mutant Ameloblastoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Baihui Miao, graduate student, Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023013
Record Dates: First submitted 2024-02-08; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Ameloblastoma
Keywords: BRAF Gene Mutation; Fenestration decompression
MeSH Terms: conditions — Ameloblastoma | interventions — dabrafenib

STUDY DESIGN:
Intervention Model Description: This study is a single-arm study that does not involve randomization or blinding, nor does it establish a parallel control group and uses external control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dabrafenib (Experimental): This study is a single-arm study that does not involve randomization or blinding, nor does it establish a parallel control group and uses external control.
  Interventions: Drug: Dabrafenib

INTERVENTIONS:
Drug: Dabrafenib — Generic name: Dabrafenib mesylate capsules Dosage form: capsule Specifications: 50mg, calculated as C23H20F3N5O2S2 Usage: Orally The dose of dabrafenib is 150 mg twice daily (equivalent to a total daily dose of 300 mg), taken at least 1 hour before or 2 hours after a meal. If you miss a dose and it is less than 6 hours before the next dose, you should not take it.
  Patients who undergo fenestrated decompression will be administered the drug for 8 weeks, with curettage performed between weeks 8 and 9. Patients undergoing curettage will continue to take dabrafenib preoperatively until a few hours before surgery, but ideally, patients will take dabrafenib within 12 hours before surgery.
  Other Names: fenestration decompression

SUMMARY:
This pilot clinical trial plans to carry out dabrafenib adjuvant therapy combined with lesion curettage after fenestrated decompressive surgery for BRAF mutation-positive multicystic ameloblastoma to explore the effectiveness of this therapy in preventing tumor recurrence, reducing or even avoiding postoperative deformity and dysfunction. effect. Based on this, we plan to launch a prospective clinical study of dabrafenib in the treatment of BRAF V600E ameloblastoma, verify the feasibility of drug treatment or drug-assisted treatment of ameloblastoma, and provide patients with a safer Effective new treatment options will benefit more patients.

DETAILED DESCRIPTION:
Main purpose:

To verify the application value of dabrafenib, a targeted drug targeting BRAF V600E mutation, combined with fenestration decompression and tumor curettage therapy in the treatment of multicystic ameloblastoma. It is expected to provide patients with a new treatment option that improves curative effect, reduces postoperative tumor recurrence, and avoids postoperative deformity.

Secondary purpose:

Study of regional heterogeneity in BRAF V600E-mutant ameloblastoma. Provide new ideas for finding other effective treatments.

Overall research design This study is a single-center, single-arm exploratory study. It is planned to enroll 10 patients with BRAF V600E mutation-positive multicystic ameloblastoma. After signing the informed consent form, you can enter the study as a subject.

Subjects will receive the study drug dabrafenib immediately after window decompression surgery. They will take dabrafenib for at least 8 weeks. Lesion curettage will be performed within the 8th to 9th week. Preoperative imaging will check the tumor volume. zoomed out situation. Patients whose lesions are not completely curettaged may choose to resume the dose of dabrafenib they received immediately before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histology confirmed ameloblastoma.
* The patient was tested positive for BRAF V600E mutation.
* Eligible patients must have evaluable lesions within the jaw that meet RECIST criteria.
* Be 18 years or older.
* Laboratory test results:

ANC > 1.5 x 109/L. PLT > 99 x 109/L. Hemoglobin >8 g/dL. Tbili < 1.6 × ULN. AST, ALT and alkaline phosphate < 2.6 times the upper limit of normal (ULN) . Serum creatinine ≤1.5 mg/dL, or serum creatinine >1.5 mg/dL, creatinine clearance must be ≥50ml/min.

PR / INR, PTT ≤ 1.3 × ULN, patients receiving anticoagulation therapy can participate in the trial if their INR is within the therapeutic range before randomization.

* Patients of childbearing potential must agree to use effective contraception for at least 6 months after treatment with dabrafenib.
* Be able to swallow and retain oral medications and must not have any clinically significant gastrointestinal abnormalities that may alter absorption, such as malabsorption syndrome or major resection of the stomach or intestines.
* The left ventricular ejection fraction is equal to or greater than normal within 1 month of enrollment.
* Voluntarily sign the informed consent form and cooperate with the treatment.

Exclusion Criteria:

* Those who have used BRAF inhibitor treatment in the past.
* Patients with invasive malignant tumors other than ameloblastoma within 3 years, excluding cancers with high cure rates, such as early cutaneous squamous cell carcinoma (T1 N0), cervical cancer, early prostate cancer, thyroid cancer, breast cancer Cancer and malignant tumors with confirmed activating RAS mutations at any time.
* Those who have had retinal vein occlusion in the past or currently.
* Those with a history of interstitial lung disease or lung inflammation.
* Those suffering from uncontrolled hypertension (systolic blood pressure > 140 mm Hg, diastolic blood pressure > 90 mm Hg, which cannot be controlled by antihypertensive treatment), heart failure or other serious medical diseases.
* Patients with previous allergic reactions caused by compounds with similar chemical or biological components to dabrafenib or trametinib.
* Concomitantly taking strong CYP3A4 or CYP2C8 inhibitors (such as ketoconazole, nefazodone, clarithromycin, gemfibrozil) or strong inducers (such as rifampicin, phenytoin, carbamazepine, phenobarbide) appropriate).
* Those who take proton pump inhibitors, H2 receptor antagonists, and antacids at the same time.
* People with known G6PD deficiency.
* Pregnant or lactating patients. Women of childbearing potential must have a negative serum pregnancy test within 14 days of enrollment. Women of childbearing potential must agree to use effective contraception 14 days before enrollment, throughout treatment, and for 4 to 6 months after the last dose of study treatment.
* Those with electrogram QTcB > 480 ms within 14 days of enrollment.
* Patients with congestive heart failure NYHA grade III or more severe (physical activity is significantly limited).
* History of acute coronary syndrome (including myocardial infarction or unstable angina), coronary angioplasty or stent implantation within 6 months, or current clinically significant uncontrolled disease recorded by echocardiography History or evidence of arrhythmias or intracardiac defibrillators or cardiac valve morphological abnormalities (≥Grade 2). Subjects with grade 1 abnormalities (ie, mild regurgitation/stenosis) are eligible for enrollment. Subjects with moderate valve thickening were not eligible. Subjects with controlled atrial fibrillation for >30 days prior to dosing were eligible.
* Patients with previous systemic anti-cancer treatment (chemotherapy, immunotherapy, biological therapy, vaccine treatment within 3 weeks before study treatment, or chemotherapy without delayed toxicity within 2 weeks before study treatment).
* Any serious or unstable pre-existing illness, mental illness, or other condition that may affect subject safety, obtaining informed consent, or compliance with research procedures.
* History of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. Subjects with laboratory evidence of cure of HBV and/or HCV will be admitted.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 2 months after fenestration decompression
  It is defined as the proportion of patients whose tumor volume has been reduced by 40% between treatment after fenestration decompression and before curettage, that is, the sum of the proportions of complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Relapse-free survival | 2 years after tumor curettage
  The time from tumor curettage to disease recurrence (local, regional or distant metastasis), whichever occurs first, is determined according to the investigator's assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Li, Principal Investigator — Shandong University School of Stomatology

IPD SHARING:
Plan to Share IPD: No